CLINICAL TRIAL: NCT04705753
Title: Evaluation of the Clinical Outcomes and the Quality of Life of Patients Exhibiting Symptoms Characteristic of Viral Respiratory Infection (VRI), Including Infection by SARS-CoV-2 (COVID-19), and Assessment of the Clinical Effectiveness of a Herbal Extract (Cretan IAMA) in These Patients and the People Cohabiting With Them Via an Open-label, Single-arm Trial
Brief Title: Assessment of the Clinical Effectiveness of a Herbal Extract (Cretan IAMA) in Patients With Viral Respiratory Infections, Including COVID-19, in Primary Healthcare Settings, and Co-assessment of Its Prophylactic Effect in People Cohabiting With These Patients
Acronym: COVID-19-IAMA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Crete (Other)
Collaborators: Galenica SA (Unknown); Olvos Science SA (Unknown)
Responsible Party: Principal Investigator, Christor Lionis, Professor of General Practice and Primary Healthcare, Director of the Clinic of Social and Family Medicine, University of Crete
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 78/26.03.2020
Record Dates: First submitted 2021-01-06; First posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Covid19; Viral Infection; Respiratory Viral Infection
Keywords: Infectious disease; Herbal Medicine; Botanical Medicine
MeSH Terms: conditions — COVID-19; Virus Diseases; Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cretan IAMA (CAPeo) (Experimental): All patients are to receive Cretan IAMA (CAPeo) from Day 1.
  Interventions: Dietary Supplement: Cretan IAMA

INTERVENTIONS:
Dietary Supplement: Cretan IAMA — Cretan IAMA (CAPeo) soft gels, 1 ml/day of a 1.5% essential oil combination from three aromatic plants (Thymbra 59 capitata (L.) Cav., Origanum dictamnus L., Salvia fruticosa Mill.) in extra virgin olive oil
  Other Names: CAPeo

SUMMARY:
This single-arm, open-label small interventional proof-of-concept (POC) study study aims:

1. to assess the clinical outcomes of patients exhibiting viral respiratory infection (VRI) symptoms and seeking primary healthcare (PHC) services at the time of the COVID-19 pandemic,
2. to assess the clinical effectiveness of the Cretan IAMA (CAPeo), a herbal extract combination, for these patients, including in terms of symptom resolution (symptom frequency, duration) and intensity), and
3. to investigate its prophylactic effect in terms of transmission prevention for people cohabiting with the patients exhibiting VRI symptoms.

DETAILED DESCRIPTION:
Cretan IAMA (CAPeo) is an essential oil mixture of three native herbs of Crete (Thymbra capitata (L.) Cav., Salvia fruticosa Mill. and Origanum dictamnus L.), which exhibits remarkable in vitro antiviral activity against Influenza A & B and the Human Rhinovirus HRV-14 strains, decreasing the symptoms of upper respiratory tract viral infections. It has also been proven safe in experimental animals and humans. There is currently a strong unmet medical need for safe and effective therapeutic regimens for patients in ambulatory settings. Given its properties, it was, therefore, deemed both appropriate and urgent to explore its potential in the context of COVID-19 for patients in primary care settings. It was also deemed important to investigate the Cretan IAMA (CAPeo) regarding prophylactic treatment for people coming in close contact with these ambulatory patients.

* Single-arm, open label (proof-of-concept) study to assess the potential of Cretan IAMA (CAPeo) benefit of COVID-19 as a therapeutic and prophylactic agent
* VRI/COVID-19 patients seeking primary health care services at home
* SARS-CoV-2 infection testing by real-time RT-PCR, performed in the regional COVID-19 reference centre (Laboratory of Clinical Virology, University of Crete, School of Medicine)
* Cretan IAMA (CAPeo) to be administered in the form of two 0.5 ml soft capsules, in a concentration of 15 ml/L, daily for two weeks (14 days), per os
* Data collection on Day 1 (baseline), Day 4, Day 7 and Day 14

ELIGIBILITY:
Inclusion Criteria:

* For the patients:

  * Any woman or man requesting a home visit and having symptoms characteristic of viral infection, with initial manifestation within the previous 48-72 hrs. Such symptoms may include sudden fever onset, accompanied by one or more of the following symptoms: dry cough, sore throat, nasal congestion, headache, musculoskeletal pain, perspiration, fatigue, malaise, blurry vision, loss of the sense of smell.
* For the people cohabiting with patients:

  * Any woman or man cohabiting with study patients.

Exclusion Criteria:

* Children and adolescents under the age of 18 years;
* Pregnant women;
* Persons suffering from a pre-existing condition preventing them from autonomously providing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Number of patients with symptom resolution | 2 weeks (14 days)
  Number of patients with symptoms recorded at baseline resolving at 2 weeks (14 days) or sooner
Number of people cohabiting with a patient not developing VRI symptoms | 2 weeks (14 days) )
  Number of people cohabiting with a patient who did not develop VRI symptoms (per patient) at 2 weeks (14 days)

SECONDARY OUTCOMES:
Median time to full symptom resolution | 2 weeks (14 days)
  Median time to full symptom resolution, including those emerging after Day 1 adjusted for symptoms emerging after Day 1 (Baseline symptoms)
Intensity of symptoms | 2 weeks (14 days)
  Intensity of symptoms, incl. of those emerging after Day 1 (Baseline symptoms), and adjusted for symptoms emerging after Day 1 (Baseline symptoms), scoring on the seven-point Likert scale based on a questionnaire adapted from the Wisconsin Upper Respiratory System Survey - A seven-point Likert scale allowed recording 131 of reported symptoms starting from 1 (minor) to 2 (very mild) and 3 (mild), 4 (somewhat moderate) and 132 5 (moderate) and culminating to 6 (severe) and 7 (very severe).
Duration of symptoms | 2 weeks (14 days)
  Duration of symptoms, incl. of those emerging after Day 1 (Baseline symptoms) and adjusted for symptoms emerging after Day 1 (Baseline symptoms)
Number of patients whose symptoms never exceeded a score of 3-4 (mild) | 2 weeks (14 days)
  Number of patients whose symptoms never exceeded a score of 3-4 (mild) on the seven-point Likert scale based on a questionnaire adapted from the Wisconsin Upper Respiratory System Survey
Quality of life (QoL) of patients | 2 weeks (14 days)
  EQ-5D-5L measurement of QoL

CONTACTS AND LOCATIONS:
Overall Officials: Christos Lionis, Principal Investigator — University of Crete
Locations (1):
- Cretan Medicare, Heraklion, Crete, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lionis C, Faresjo A, Skoula M, Kapsokefalou M, Faresjo T. Antioxidant effects of herbs in Crete. Lancet. 1998 Dec 19-26;352(9145):1987-8. doi: 10.1016/S0140-6736(05)61333-5. No abstract available. PMID 9872255
- [Result] Duijker G, Bertsias A, Symvoulakis EK, Moschandreas J, Malliaraki N, Derdas SP, Tsikalas GK, Katerinopoulos HE, Pirintsos SA, Sourvinos G, Castanas E, Lionis C. Reporting effectiveness of an extract of three traditional Cretan herbs on upper respiratory tract infection: results from a double-blind randomized controlled trial. J Ethnopharmacol. 2015 Apr 2;163:157-66. doi: 10.1016/j.jep.2015.01.030. Epub 2015 Jan 30. PMID 25645191
- [Result] Tseliou, M., Pirintsos, S. A., Lionis, C., Castanas, E., and Sourvinos, G. (2019). Antiviral effect of an essential oil combination derived from three aromatic plants (Coridothymus capitatus (L.) Rchb. f., Origanum dictamnus L. and Salvia fruticosa Mill.) against viruses causing infections of the upper respiratory tract. J. Herb. Med. 17-18, 100288. doi:10.1016/j.hermed.2019.100288.
- [Result] Pirintsos SA, Bariotakis M, Kampa M, Sourvinos G, Lionis C, Castanas E. The Therapeutic Potential of the Essential Oil of Thymbra capitata (L.) Cav., Origanum dictamnus L. and Salvia fruticosa Mill. And a Case of Plant-Based Pharmaceutical Development. Front Pharmacol. 2020 Nov 24;11:522213. doi: 10.3389/fphar.2020.522213. eCollection 2020. PMID 33390932
- [Result] Anastasaki M, Bertsias A, Pirintsos SA, Castanas E, Lionis C. Post-market outcome of an extract of traditional Cretan herbs on upper respiratory tract infections: a pragmatic, prospective observational study. BMC Complement Altern Med. 2017 Sep 21;17(1):466. doi: 10.1186/s12906-017-1978-7. PMID 28934952